CLINICAL TRIAL: NCT01337336
Title: Chronic Obstructive Pulmonary Disease (COPD)-Related Outcomes and Costs for Patients on Combination Fluticasone Propionate-Salmeterol Xinafoate 250/50mcg Versus Anticholinergics in a Comorbid COPD-Depression/Anxiety Population
Brief Title: Chronic Obstructive Pulmonary Disease (COPD)-Related Outcomes and Costs for Patients on Combination Fluticasone Propionate-Salmeterol Xinafoate 250/50mcg Versus Anticholinergics in a COPD-Comorbid Depression/Anxiety Population
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113902
Record Dates: First submitted 2011-04-15; First posted 2011-04-18 (Estimated); Results first posted 2011-05-20 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone-Salmeterol Drug Combination; Cholinergic Antagonists; Tiotropium Bromide; Ipratropium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- COPD patients with comorbid depression/anxiety: Patients aged 40 and over with COPD and comorbid depression/anxiety. Managed care enrolees (aged >40 years) having newly initiated drug therapy with FSC or AC during the identification period (01/01/2004 to 06/30/2008) to treat COPD with a medical or pharmacy claim for depression before and 60 days post index date were the target population. The first fill date of FSC or AC was the index date.
  Interventions: Drug: fluticasone propionate/salmeterol xinafoate; Drug: Anticholinergics

INTERVENTIONS:
Drug: fluticasone propionate/salmeterol xinafoate — combination fluticasone priopionate and salmeterol xinafoate 250/50mcg
  Other Names: FSC; Advair (TM)
Drug: Anticholinergics — tiotropium; ipratropium alone; or ipratropium + albuterol
  Other Names: tiotropium; ACs; ipratropium

SUMMARY:
The objective of this study was to examine COPD-related outcomes for patients with comorbid depression/anxiety who are on combination fluticasone propionate/salmeterol xinafoate compared to those receiving anticholinergics.

The prevalence of comorbid depression/anxiety in patients with chronic obstructive pulmonary disease (COPD) is estimated to be high and range from 10-40%, given that the risk of depression/anxiety symptoms is almost 3 times higher in patients with versus without COPD. Additionally, patients with comorbid COPD and depression/anxiety have higher COPD-related healthcare utilization and costs compared to those without depression/anxiety. Therapy with maintenance medications for COPD has been recommended to prevent future adverse COPD outcomes, but the impact of initiating these interventions has not yet been evaluated in a higher-risk population with comorbid COPD-depression/anxiety. The present study compares the risk of COPD exacerbations and COPD-related costs in patients initiating maintenance medications for treatment of COPD in a comorbid COPD/depression-anxiety population. Maintenance medications include inhaled corticosteroid (ICS), long-acting beta agonist (LABA), combination drug product of ICS+LABA, and anti-cholinergics (AC) including tiotropium (TIO) and ipratropium or combination ipratropium-albuterol (collectively abbreviated as IPR).

DETAILED DESCRIPTION:
This was a retrospective cohort study using a large administrative database (study period: 1/1/2003 through 6/30/2009). Date of first FSC or ACs (tiotropium; ipratropium alone or in combination with albuterol) was defined as the index date. Managed care enrollees (aged >40 years) having at least one medical claim with a primary diagnosis of COPD (ICD code 491.xx, 492.xx and 496.xx) and a diagnosis of depression (at least one claim with depression/anxiety or at least one prescription claim for depression/anxiety) in one-year pre-index and within 60-days post-index were defined in the comorbid population. Patients were continuously eligible throughout the one-year pre and post-index periods. Negative binomial models were used to analyze number of COPD-related events [hospitalization (IP), emergency department (ED), office visits with oral steroid and/or antibiotic prescription within 5 days (OV+Rx)] and logistic regression was used to examine risk of COPD events between the two cohorts. COPD-related costs were compared between the two cohorts using - generalized linear model with log-link/gamma distribution after adjusting for baseline differences.

Specifically the study hypothesis for the primary outcome being tested was:

Ho: There is no difference in risk of any COPD-related exacerbation between FSC and AC cohorts Ha: There is a difference in risk of any COPD-related exacerbation between FSC and AC cohorts

Hypothesis for the key secondary outcome of COPD-related costs that was tested was:

Ho: There is no difference in COPD-related costs between FSC and AC cohorts Ha: There is a difference in COPD-related costs between FSC and AC cohorts

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD in any field in the pre-index period and 60 days after the index date
* Diagnosis of depression/anxiety in any field and a medication for treating depression/anxiety in the pre-index period and 60 days after the index date
* Index date occurs during identification period
* Patients must be continuously eligible during 1-year pre and 1-year post-index date and be of at least 40 years of age

Exclusion Criteria:

* comorbid conditions (respiratory cancer, cystic fibrosis, fibrosis due to tuberculosis, and bronchiectasis, pneumonociosis, pulmonary fibrosis, pulmonary tuberculosis, sarcoidosis) during the 1 year pre or post-index periods
* No other maintenance medications other than the index medication on or 60 days after the index date

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population included patients with both COPD and depression/anxiety. They were identified as follows: Patients who had at least one pharmacy claim for a maintenance medication used to treat COPD were identified. Of these, patients were considered to have comorbid depression/anxiety if they had at least one prescription claim for a medication used to treat depression/anxiety and a diagnosis code for depression/anxiety during 1 year pre-index or within 60 days after the index date.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2010-10; Primary Completion 2010-11 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Groups:
- FSC Cohort: Fluticasone/Salmeterol Combination (FSC) 250/50 micrograms (mcg) twice a day
- AC Cohort: Anticholinergics (AC) include Tiotropium, Ipratropium, and Ipratropium-albuterol combination drug product. Due to the retrospective nature of this study, dosing information is not available.
Period: Overall Study
Arm/Group | FSC Cohort | AC Cohort
Started | 1078 | 2923
Completed | 1078 | 2923
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FSC Cohort | AC Cohort | Total
Number analyzed (Participants) | 1078 | 2923 | 4001
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.8 (9.8) | 60.3 (10.3) | 59.6 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 742 | 1910 | 2652
  Male | 336 | 1013 | 1349

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Chronic Obstructive Pulmonary Disease (COPD)-Related Exacerbation
Description: The number of participants with any of the following COPD-related exacerbations during the follow-up period was computed: COPD-related hospitalization, emergency room (ER) visit, or physician visit with a prescription (Rx) for oral corticosteroid (OCS) or antibiotic within 5 days of the visit. The index date is defined as the date of first chronologically occurring COPD maintenance medication of interest during an identification period spanning January 1, 2004 to June 30, 2008.
Time Frame: Maximum of 1 year after index date (January 1, 2004 to June 30, 2009)
Population: Managed care enrollees (aged >=40 years) diagnosed with COPD (ICD code 491.xx, 492.xx, and 496.xx) and depression/anxiety before or within 60 days of the date of first prescription for a maintenance medication for COPD (index date).
Measure: Number; unit: participants
Arm/Group | FSC Cohort | AC Cohort
Number analyzed (Participants) | 1078 | 2923
participants | 200 | 674
Statistical Analysis 1: Comparison: FSC Cohort vs AC Cohort; Test type: Superiority or Other; p = 0.002, Chi-squared; Odds Ratio (OR) = 1.30, 95% CI [1.08 to 1.56] — Estimated value obtained from logistic regression model controlling for differences between cohorts at baseline on demographic variables, proxy measures of COPD severity, and measures of overall disease burden

2. Secondary Outcome: Number of Participants With the Indicated COPD-related Exacerbations
Description: The number of participants with a COPD-related exacerbation was identified during the follow-up period. Four types of COPD-related exacerbations were defined: COPD-related hospitalization, ER visit, physician visit with a prescription (Rx) for oral corticosteroid or antibiotic within 5 days of the visit, or combined occurrence of COPD-related hospitalization/ER visit. The index date is defined as the date of first chronologically occurring COPD maintenance medication of interest during an identification period spanning January 1, 2004 to June 30, 2008.
Time Frame: Maximum of 1 year after index date (January 1, 2004 through June 30, 2009)
Population: Managed care enrollees (aged >=40 years) diagnosed with COPD (ICD code 491.xx, 492.xx, and 496.xx) and depression/anxiety before or within 60 days of the date of first prescription for a maintanance medication for COPD (index date).
Measure: Number; unit: participants
Arm/Group | FSC Cohort | AC Cohort
Number analyzed (Participants) | 1078 | 2923
participants
  COPD-related hospitalization | 35 | 168
  COPD-related ER visit | 37 | 171
  COPD-related physician + Rx visit | 156 | 448
  COPD-related hospitalization/ER visit | 63 | 307
Statistical Analysis 1: Comparison: FSC Cohort vs AC Cohort; Test type: Superiority or Other; p = 0.002, Chi-squared — COPD-related hospitalization; Odds Ratio (OR) = 1.56, 95% CI [1.02 to 2.38] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: FSC Cohort vs AC Cohort; Test type: Superiority or Other; p = 0.002, Chi-squared — COPD-related ER visit; Odds Ratio (OR) = 1.65, 95% CI [1.14 to 2.39] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: FSC Cohort vs AC Cohort; Test type: Superiority or Other; p = 0.503, Chi-squared; COPD-related physician + Rx visit; Odds Ratio (OR) = 1.14, 95% CI [0.93 to 1.40] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: FSC Cohort vs AC Cohort; Test type: Superiority or Other; p < 0.001, Chi-squared; COPD-related hospitalization/ER visit; Odds Ratio (OR) = 1.71, 95% CI [1.26 to 2.31] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Mean Annual COPD-related Costs Per Participant
Description: Cost categories included medical, pharmacy, and total (calculated as the sum of medical and pharmacy). COPD-related medical costs were computed using claims with a primary diagnosis of COPD, and COPD-related pharmacy costs were computed using the paid amounts of pharmacy claims for prescription medication used for COPD.The index date is defined as the date of first chronologically occurring COPD maintenance medication of interest during an identification period spanning January 1, 2004 to June 30, 2008.
Time Frame: Maximum of 1 year after index date (January 1, 2004 through June 30, 2009)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: United States (US) dollars
Arm/Group | FSC Cohort | AC Cohort
Number analyzed (Participants) | 1078 | 2923
United States (US) dollars
  COPD-related total costs | 1604 (3187) | 1687 (4299)
  COPD-related pharmacy costs | 934 (814) | 684 (724)
  COPD-related medical costs | 670 (2923) | 1003 (4095)

4. Secondary Outcome: Number of the Indicated COPD-related Exacerbations
Description: The number of COPD-related exacerbations was identified during the follow-up period. Five types of COPD-related exacerbations were defined: -COPD-related hospitalization, ER visit, physician visit with a prescription (Rx) for oral corticosteroid or antibiotic within 5 days of the visit, combined occurrence of COPD-related hospitalization/ER visit, or combined occurrence of any COPD-related exacerbation. The index date is defined as the date of first chronologically occurring COPD maintenance medication of interest during an identification period spanning January 1, 2004 to June 30, 2008.
Time Frame: Maximum of 1 year after index date (January 1, 2004 through June 30, 2009)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of exacerbations
Arm/Group | FSC Cohort | AC Cohort
Number analyzed (Participants) | 1078 | 2923
number of exacerbations
  COPD-related hospitalization | 0.04 (0.2) | 0.07 (0.3)
  COPD-related ER visit | 0.06 (0.4) | 0.07 (0.4)
  COPD-related physician (phy)+Rx visit | 0.19 (0.6) | 0.20 (0.6)
  COPD-related hospitalization/ER visit | 0.09 (0.5) | 0.14 (0.5)
  COPD-related hospitalization/ER visit/phy+Rx visit | 0.29 (0.8) | 0.34 (0.8)
Statistical Analysis 1: Comparison: FSC Cohort vs AC Cohort; Test type: Superiority or Other; p = 0.0004, t-test, 2 sided — COPD-related hospitalization; Incident Rate Ratio = 1.46, 95% CI [1.01 to 2.09] — Estimated value obtained from zero-inflated negative binomial model controlling for differences between cohorts at baseline on demographic variables, proxy measures of COPD severity, and measures of overall disease burden
Statistical Analysis 2: Comparison: FSC Cohort vs AC Cohort; Test type: Superiority or Other; p = 0.208, t-test, 2 sided — COPD-related ER visit; Incident Rate Ratio = 1.27, 95% CI [0.89 to 1.82] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: FSC Cohort vs AC Cohort; Test type: Superiority or Other; p = 0.671, t-test, 2 sided — COPD-related physician + Rx visit; Incident Rate Ratio = 1.09, 95% CI [0.90 to 1.32] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: FSC Cohort vs AC Cohort; Test type: Superiority or Other; p = 0.009, t-test, 2 sided — COPD-related hospitalization/ER visit; Incident Rate Ratio = 1.31, 95% CI [1.05 to 1.72] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: FSC Cohort vs AC Cohort; Test type: Superiority or Other; p = 0.052, t-test, 2 sided — COPD-related hospitalization/ER visit/physician + Rx visit; Incident Rate Ratio = 1.16, 95% CI [0.98 to 1.37] — [estimate comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Description: This study was a retrospective observational study; thus, no serious adverse events or adverse events were collected.
Groups:
- AC Cohort: Anticholinergics (AC) include iotropium, and Ipratropium, Ipratropium-albuterol combination drug product. Due to the retrospective nature of this study, dosing information is not available.
Arm/Group | FSC Cohort | AC Cohort
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.